CLINICAL TRIAL: NCT04802083
Title: SOLIRIS® (Eculizumab) for the Treatment of Participants With Coronavirus Disease 2019 (COVID-19) - An Expanded Access Protocol
Brief Title: COVID-19 Soliris Expanded Access Protocol
Status: No longer available | Type: Expanded Access
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ECU-COV-402
Record Dates: First submitted 2021-02-17; First posted 2021-03-17 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Covid19
Keywords: Soliris; eculizumab; C5 inhibitor; COVID-19; SARS-COV-2; acute lung injury; severe pneumonia; acute respiratory distress syndrome; severe acute respiratory syndrome coronavirus 2; severe acute respiratory syndrome; multi-organ injury; hospitalization; antibodies, monoclonal, humanized; emergency treatment; viral; expanded access
MeSH Terms: conditions — COVID-19; Acute Lung Injury; Pneumonia; Respiratory Distress Syndrome; Severe Acute Respiratory Syndrome | interventions — eculizumab; Antibodies, Monoclonal

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: Eculizumab — Eculizumab 900-1200 mg will be administered intravenously.
  Other Names: Soliris, monoclonal antibody

SUMMARY:
This protocol provides participants with COVID-19 access to Soliris.

DETAILED DESCRIPTION:
This is an open-label, multicenter, expanded access protocol that will provide access to Soliris for participants diagnosed with severe acute respiratory syndrome coronavirus 2 (SARS-COV-2) infection with a clinical presentation consistent with COVID-19 associated organ injury, such as acute respiratory distress syndrome, stroke, or acute renal failure. Participants who qualify for emergency treatment (whether in an inpatient or outpatient setting) will be offered the opportunity to receive up to 7 infusions of Soliris over approximately 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 18 years of age and body weight ≥ 40 kg.
2. Confirmed diagnosis of SARS-COV-2 infection by any method used by the institution (eg, via reverse transcriptase polymerase chain reaction and/or antibody test).
3. Willing to receive vaccination against Neisseria meningitidis and prophylactic antibiotics against meningococcal infections if the participant has not been vaccinated within 5 years prior to Day 1.
4. In the opinion of the Investigator, the participant is suitable to be enrolled in the expanded access protocol (EAP), based on the participant's overall clinical condition and the known Soliris benefit/risk profile.

Exclusion Criteria:

1. Unresolved Neisseria meningitidis infection.
2. Known hypersensitivity to murine proteins or to an excipient of Soliris.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult